CLINICAL TRIAL: NCT06904716
Title: The Study of Transcranial Magnetic Stimulation in the Regulation of Spinocerebellar Ataxia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Fei Xiao, Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-140
Record Dates: First submitted 2025-03-11; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Spinocerebellar Ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Perform low-frequency Transcranial Magnetic Stimulation (TMS) on the left and right cerebellar hemispheres and the vermis of the cerebellum, twice a day for a total of 7 days.
  Interventions: Other: Transcranial magnetic stimulation
- Controls (No Intervention): The healthy control group does not receive any intervention.

INTERVENTIONS:
Other: Transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation
  Arms: Test group

SUMMARY:
Spinocerebellar ataxia (SCA) is a group of hereditary neurological diseases caused by gene mutations leading to degenerative changes in the cerebellum, brainstem, and spinal cord. A key pathogenic mechanism of SCA is the repeated expansion of cytosine - adenine - guanine (CAG) trinucleotides in the coding region of specific genes. These repeated expansions are translated into abnormally large polyglutamine (PolyQ) tracts in proteins. These polyglutamine (PolyQ) tracts can cause changes in the excitability of the cerebral cortex in SCA patients. Quantitative electroencephalogram analysis (qEEG) is a modern type of electroencephalogram analysis that uses complex mathematical algorithms to process, transform, and analyze EEG signals, bringing new technologies for EEG signal feature extraction: specific frequency band and signal complexity analysis, connectivity analysis, and network analysis. It is sensitive to early neurodegenerative lesions. Using spectral analysis, nonlinear dynamics analysis, and functional connectivity analysis, we can explore the changes in cortical excitability and abnormal brain networks in SCA patients. Currently, the exploration of the quantitative electroencephalogram characteristics of SCA patients is still insufficient.

ELIGIBILITY:
Inclusion Criteria:

1. Spinocerebellar ataxia patients confirmed through genetic testing
2. Patient aged 18-75
3. Patients who can walk independently (with the aid of a cane/walker) without assistance from others.
4. The SARA score exceeds 3.

Exclusion Criteria:

1. Patients with unstable neurological disorders or accompanying medical conditions (such as stroke, arthritis, etc.)
2. Patients with significantly abnormal clinical indicators identified during screening
3. Patients concurrently participating in another clinical study
4. Patients with untreated intracranial hypertension, depression, dementia, or psychiatric disorders
5. Patients with severe heart disease
6. Patients who are wheelchair users
7. pregnant woman
8. Patients who cannot establish their identity or have limited legal capacity
9. Patients with contraindications for rTMS, including metallic objects in the head, history of neurosurgery, ferromagnetic bioimplants, metal coatings, history of seizures, autism, current use of protease inhibitors or other medications that may increase the risk of rTMS-induced seizures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia | Baseline and one week post-baseline (after treatment)
  The Scale for the Assessment and Rating of Ataxia (SARA) is a clinical tool used to assess the severity of ataxia. The total score range of the SARA scale is 0 to 40 points, with higher scores indicating more severe ataxia symptoms.
Resting - state electroencephalogram | baseline and one week post-baseline (after treatment)
  Use electroencephalogram (EEG) to collect the electroencephalogram data of participants with their eyes closed and in a waking state.Using spectral analysis, nonlinear dynamics analysis, and functional connectivity analysis, we can explore the changes in cortical excitability and abnormal brain networks in SCA patients.
Transcranial Magnetic Stimulation - Electroencephalogram（TMS-EEG） | Baseline and one week post-baseline (after treatment)
  Transcranial magnetic stimulation is utilized to stimulate the brain, and then EEG data is immediately collected from participants using EEG to collect closed-eye, awake EEG data.Using time-frequency analysis, nonlinear dynamics analysis, and functional connectivity analysis, we can explore the changes in cortical excitability and abnormal brain networks in SCA patients.

SECONDARY OUTCOMES:
The International Cooperative Ataxia Rating Scale (ICARS) | Baseline and one week post-baseline (after treatment)
  The International Cooperative Ataxia Rating Scale (ICARS) is a widely used clinical tool designed to assess the severity of ataxia, particularly in patients with cerebellar disorders. The total score range of the ICARS scale is 0 to 100 points, with higher scores indicating more severe ataxia symptoms.
The Neurological Examination Score for the assessment of Spinocerebellar Ataxias (NESSCA) | Baseline and one week post-baseline (after treatment)
  The Neurological Examination Score for the Assessment of Spinocerebellar Ataxias (NESSCA) is a clinical tool specifically designed to evaluate the severity of spinocerebellar ataxias (SCAs).The total score range of the NESSCA scale is 0 to 60 points, with higher scores indicating more severe ataxia symptoms.
The EQ Visual Analogue Scale | Baseline and one week post-baseline (after treatment)
  The EQ Visual Analogue Scale (EQ-VAS) is a component of the EuroQol Five Dimensions Questionnaire (EQ-5D) used to assess a patient's subjective perception of their overall health.The EQ-VAS ranges from 0 to 100. 0: Represents "the worst imaginable health state." 100: Represents "the worst imaginable health state." High scores (closer to 100): Indicate that the patient perceives their health as very good.Low scores (closer to 0): Indicate that the patient perceives their health as very poor.
Gait analysis | Baseline and one week post-baseline (after treatment)
  The researchers use gait sensors to collect gait data

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliatted Hospital of Chongqing medical Uiversity, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
With the consent of both researchers and participants, the original data can be obtained by contacting with the corresponding member.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2023.05~2025.05
Access Criteria: After obtaining informed consent from the patients and ensuring compliance with ethical principles, this study uses Case Report Forms (CRF) and questionnaires to collect subject information. The CRFs and questionnaires are stored in both paper and electronic databases. Data collection occurs after obtaining patients' informed consent at the time of their participation in the study assessment. Two members of the research team independently enter CRF data into the electronic database, and any discrepancies are reconciled before making changes to the entry. Original paper and electronic data are registered and stored in our department's clinical trial archive cabinet.